CLINICAL TRIAL: NCT07030153
Title: Genetic Variants and Their Association With Myopia Risk, Progression, and Optimal Interventions in Children
Brief Title: Association of Genetic Variants With Myopia
Status: Recruiting | Type: Observational
Sponsor: Beijing Visionly Plus Eye Hospital (Other)
Collaborators: Beijing New Vision Eye Hospital (Unknown); High Myopia Control Alliance (HIMALAYA) (Unknown)
Responsible Party: Sponsor
Other Study IDs: Precvision202501
Record Dates: First submitted 2025-04-22; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Myopia
Keywords: Myopia; genetic; intervention
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Oral swab DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Genetic and myopia onset: Identify genetic variants (GWAS/WES) associated with:
  * Myopia onset risk (high-risk SNPs ).
  * Myopia progression rate (e.g., axial elongation/year).
  Interventions: Genetic: Oral swab DNA analyzed for myopia-related gene variants
- Genetic and myopia intervention: Evaluate gene-intervention interactions for:
  * Low-dose atropine (0.01%, 0.05%).
  * Orthokeratology.
  * Defocus-incorporated spectacles.
  * Outdoor/sunlight exposure (≥2 hours/day).
  Interventions: Genetic: Oral swab DNA analyzed for myopia-related gene variants

INTERVENTIONS:
Genetic: Oral swab DNA analyzed for myopia-related gene variants — Beyond detecting links between gene variants and myopia development, the testing analyzes how these variants influence treatment effectiveness. The aim is to enable early risk prediction and personalized treatment guidance for children through oral DNA testing.

SUMMARY:
This study aims to identify genetic factors linked to myopia, including those that influence a person's risk of developing it and how quickly it progresses (like changes in eye length). It will also examine how different treatments-such as low-dose atropine drops, orthokeratology lenses, specialized glasses, and increased outdoor time-interact with these genes. Finally, the research will develop a genetic risk score to help tailor personalized myopia prevention and treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-18 years.
* Any Spherical equivalent refraction (SER)
* Parental consent for genetic testing.

Exclusion Criteria:

* Suspected genetic syndromes (e.g., Stickler, Marfan).
* Other eye diseases (e.g., glaucoma, cataracts, retinal abnormalities, strabismus).
* Prior refractive surgery

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Not limited to any specific population group
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Polygenic Risk Score (PRS) for Myopia Progression | Every 6 months for 3 years
  1. Measure the Myopia Progression Rate (Change in Diopters/year)
     * Measurement Tool: Autorefractor (Topcon KR-8900)
     * Method: Spherical equivalent refraction (SER) will be measured at baseline and every 6 months, with the annual rate of change (ΔD/year) calculated.
     * Unit: Diopters (D)
  2. Measure the Axial Length Growth Rate (mm/year)
     * Measurement Tool: Optical Biometer (Zeiss IOLMaster 700)
     * Method: Axial length (AL) will be measured at baseline and every 6 months, with the annual rate of change (Δmm/year) calcu
  3. Genetic Risk Assessment Model
     * Measurement Tool: Candidate genetic loci will be screened using whole-exome sequencing (WES)or genome-wide association study (GWAS).
     * A PRS model for myopia progression will be constructed by integrating refractive error (SER) and axial length changes using LASSO, DBSLMM or LDpred2 regression.
     * The correlation between PRS and myopia progression rate will be evaluated (R² or AUC curve).

SECONDARY OUTCOMES:
Genotype-Guided Decision Tree for Myopia Control Interventions | Every 6 months for 3 years
  1. Data Collection
     * error (spherical equivalent, ΔD/year) - Measured via autorefractor (per Primary Outcome Measure)
     * Axial length (Δmm/year) - Measured via optical biometer (per Secondary Outcome Measure)
     * Genetic Data: Myopia-associated SNPs (derived from WES/GWAS)
     * Clinical Intervention Data: Type of myopia control intervention (e.g., 0.01% atropine, orthokeratology, defocus-incorporated spectacles, myopia-control soft contact lenses)
  2. Analytical Pipeline
     * Compute individual PRS by aggregating weighted risk alleles (SNP effect sizes from GWAS or WES)
     * Optimal Intervention Stratification
     * Apply logistic regression/decision tree analysis to:Identify PRS threshold(s) predictive of treatment response. Test hypotheses ( "Subjects with PRS >X exhibit superior efficacy with atropine vs. orthokeratology")
  3. Clinical Translation
     * Generate decision trees or nomograms to visualize:
     * PRS-guided intervention selection
     * Predicted treatment efficacy probabilities

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing New Vision Eye Hospital, Beijing
  - Beijing Visionly Plus Eye Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided